CLINICAL TRIAL: NCT06709209
Title: A Novel Simplified Endoscopic Score aiMed at Evaluating Ulcerative cOlitis Activity Through TXI, RDI and NBI Vascular Assessment and at prEdicting Clinical Outcome and Its Applicability in an arTificial Intelligence System: the MONET Study
Brief Title: AI-driven Narrow-band Imaging Score for Disease Assessment and Outcome Prediction in Ulcerative Colitis
Acronym: MONET
Status: Recruiting | Type: Observational
Sponsor: University College Cork (Other)
Collaborators: Olympus (Industry)
Responsible Party: Sponsor
Other Study IDs: APC193
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Ulcerative Colitis (UC)
Keywords: Ulcerative Colitis; Virtual Chromoendoscopy; Artificial Intelligence; Disease Assessment; Outcome Prediction
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Blood Specimen Collection; Defecation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Intestinal biopsies, Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ulcerative Colitis patients: UC patients who have been scheduled for colonoscopy for disease assessment or surveillance
  Interventions: Procedure: Colonoscopy after bowel cleansing; Procedure: Intestinal biopsies; Diagnostic Test: blood sampling; Diagnostic Test: Stool; Other: Clinical follow-up

INTERVENTIONS:
Procedure: Colonoscopy after bowel cleansing — Colonoscopy will be performed using HD-WLE; TXI; RDI and NBI.
Procedure: Intestinal biopsies — During colonoscopy, at least 2 biopsies from each segment will be taken as standard of care to assess inflammation in UC
Diagnostic Test: blood sampling — Blood samples will be taken for standard of care by appropriately trained members of the clinical research team. The results of the standard of care blood will be used in the research.
Diagnostic Test: Stool — The stool sample will be sent to the laboratory for Faecal Calprotectin (FCP) as a marker of disease activity.
Other: Clinical follow-up — Patients will be followed-up at 6 and 12 months after index endoscopy. Patients will be evaluated in clinic or by telephone call and the disease will be reassessed. Partial Mayo Score (PMS) and occurrence of clinical outcomes will be evaluated.

SUMMARY:
This international multicentre prospective study aims to develop a new simple score using enhanced endoscopic techniques which focus on the vascular features of the colon and reliably distinguish between a quiescent and a mild inflammation in ulcerative colitis (UC). The diagnostic performance of the new score in defining disease activity/remission compared to existing endoscopic and histological scores and predict long-term clinical outcomes will be evaluated. The study also aims to adapt current artificial intelligence (AI) algorithms for enhanced endoscopic techniques to improve standardization in UC disease assessment and outcome prediction.

DETAILED DESCRIPTION:
This is a multicentre prospective international study. This study aims at developing a new simple endoscopic score using white light endoscopy - high definition (WLE-HD), Texture and colour enhancement imaging (TXI), red dichromatic imaging (RDI) and narrow-band imaging (NBI) modes, focusing on vascular features to distinguish between quiescent versus patchy mild Ulcerative Colitis. It will evaluate the new score's diagnostic performance in defining disease activity/remission compared to existing endoscopic and histological scores and predict long-term clinical outcomes. Finally, it also aims to develop and adapt existing artificial intelligence (AI) algorithms according to WLE-HD, TXI, RDI and NBI to grade and standardize endoscopic and histological disease assessment and predict long-term clinical outcomes.

The study will be divided in several phases:

* In the first phase, the score will be developed on the first 30 consecutive virtual electronic chromoendoscopy (VCE) videos (using TXI-RDI and NBI) of UC patients, with different grade of disease activity. Experts in inflammatory bowel disease (IBD) endoscopy will review images and videos from recruited patients to define the endoscopic mucosal and vascular features of the new score. These will be used for a stepwise discussion. A round table discussion using modified Delphi method will be conducted by experts worldwide to ensure equal participation and identify the best component descriptors of endoscopic vascular healing. The components that will achieve 100% consensus will be selected, and the most important endoscopy predictive variables will be confirmed by using a machine learning technique. Finally, a new endoscopic score will be generated. This should be reproducible, valid and responsive.
* In the second phase, the new endoscopic scoring system will be validated in a large cohort of UC patients, focusing on patients with quiescent disease versus patchy mild colitis. Diagnostic accuracy, interobserver agreement and ability to predict clinical outcome according to the new endoscopic score focused on vascular features assessed with VCE will be evaluated
* In the third phase, the reproducibility of the new endoscopic scoring system will be evaluated among gastroenterologists with different levels of experience through a short survey and a computerised training module.
* In the fourth phase, new and existing AI algorithms will be developed and adapted to these endoscopic videos and histological images to grade and standardize endoscopic and histological disease assessment and predict long-term clinical outcome in UC.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 to 75 years old
* Established diagnosis of UC (for at least six months in duration), independently from their active treatment
* Undergoing endoscopy for disease activity assessment or cancer surveillance.

Exclusion Criteria:

* Contraindications to endoscopy (including toxic megacolon) and biopsies (including severe coagulopathy/thrombocytopenia)
* Poor bowel preparation (defined as total BBPS <6 or BBPS <2 in observed segment for sigmoidoscopy)
* Significant co-morbidities limiting life expectancy and conferring high risk of endoscopy
* Pregnant and breast-feeding subjects
* Inability to provide informed consent
* If the participant has been in a recent experimental trial, these must have been completed not less than thirty days prior to this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females between 18 and 75 years old with an established diagnosis of UC, who have undergone colonoscopy for disease assessment and surveillance will be consecutively recruited after obtaining written consent. The sample size in 300.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of the new scoring system | 6 months
  To evaluate the diagnostic performance of the new score in evaluating endoscopic and histological activity

SECONDARY OUTCOMES:
Correlation with existing score | 2 years
  To evaluate the new score's diagnostic performance in defining disease activity/remission compared to existing endoscopic and histological scores and predict long-term clinical outcomes
AI development | 2 years
  Develop and adapt existing AI algorithms according to WLE-HD, TXI, RDI and NBI to grade and standardize endoscopic and histological disease assessment and predict long-term clinical outcomes in UC

CONTACTS AND LOCATIONS:
Overall Officials: Marietta Iacucci, MD, Principal Investigator — University College Cork
Locations (11):
- University of Leuven, Leuven, Belgium
- Klinikum Luneburg, Lüneburg, Germany
- University College Cork, Cork, Co Cork, Ireland
- Italy (6):
  - Ospedale S. Maria del Prato, Feltre, Belluno
  - University of Bari, Bari
  - Istituto Clinico Humanitas, Milan
  - University Vita-Salute San Raffaele, Milan
  - University of Naples, Naples
  - University of Pavia, Pavia
- Showa University, Tokyo, Japan
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rath T, Atreya R, Bodenschatz J, Uter W, Geppert CE, Vitali F, Fischer S, Waldner MJ, Colombel JF, Hartmann A, Neurath MF. Intestinal Barrier Healing Is Superior to Endoscopic and Histologic Remission for Predicting Major Adverse Outcomes in Inflammatory Bowel Disease: The Prospective ERIca Trial. Gastroenterology. 2023 Feb;164(2):241-255. doi: 10.1053/j.gastro.2022.10.014. Epub 2022 Oct 21. PMID 36279923
- [Background] Iacucci M, Cannatelli R, Parigi TL, Nardone OM, Tontini GE, Labarile N, Buda A, Rimondi A, Bazarova A, Bisschops R, Del Amor R, Meseguer P, Naranjo V, Ghosh S, Grisan E; PICaSSO group. A virtual chromoendoscopy artificial intelligence system to detect endoscopic and histologic activity/remission and predict clinical outcomes in ulcerative colitis. Endoscopy. 2023 Apr;55(4):332-341. doi: 10.1055/a-1960-3645. Epub 2022 Oct 13. PMID 36228649
- [Background] Hashimoto Y, Kuribayashi S, Sato K, Itoi Y, Nakata K, Kasuga K, Tanaka H, Hosaka H, Ikota H, Iacucci M, Uraoka T. Validation of red dichromatic imaging score (RDI score) to evaluate the severity of ulcerative colitis. Surg Endosc. 2023 May;37(5):3627-3633. doi: 10.1007/s00464-022-09852-0. Epub 2023 Jan 10. PMID 36627537
- [Background] Iacucci M, Smith SCL, Bazarova A, Shivaji UN, Bhandari P, Cannatelli R, Daperno M, Ferraz J, Goetz M, Gui X, Hayee B, De Hertogh G, Lazarev M, Li J, Nardone OM, Parra-Blanco A, Pastorelli L, Panaccione R, Occhipinti V, Rath T, Tontini GE, Vieth M, Villanacci V, Zardo D, Bisschops R, Kiesslich R, Ghosh S. An International Multicenter Real-Life Prospective Study of Electronic Chromoendoscopy Score PICaSSO in Ulcerative Colitis. Gastroenterology. 2021 Apr;160(5):1558-1569.e8. doi: 10.1053/j.gastro.2020.12.024. Epub 2021 Feb 6. PMID 33347880
- [Background] Sasanuma S, Ohtsuka K, Kudo SE, Ogata N, Maeda Y, Misawa M, Mori Y, Kudo T, Hisayuki T, Wakamura K, Hayashi T, Katagiri A, Miyachi H, Baba T, Ishida F. Narrow band imaging efficiency in evaluation of mucosal healing/relapse of ulcerative colitis. Endosc Int Open. 2018 May;6(5):E518-E523. doi: 10.1055/s-0044-102297. Epub 2018 Apr 18. PMID 29713677
- [Background] He T, Zong L, Pan P, Sun S, Qu H. Predicting Histological Healing and Recurrence in Ulcerative Colitis by Assessing Mucosal Vascular Pattern Under Narrow-Band Imaging Endoscopy. Front Med (Lausanne). 2022 Jun 30;9:869981. doi: 10.3389/fmed.2022.869981. eCollection 2022. PMID 35847771
- [Background] Hayashi Y, Takabayashi K, Kato M, Tojo A, Aoki Y, Hagihara Y, Yoshida K, Yoshimatsu Y, Kiyohara H, Sugimoto S, Nanki K, Mikami Y, Sujino T, Mutaguchi M, Kawaguchi T, Hosoe N, Yahagi N, Ogata H, Kanai T. Usefulness of texture and color enhancement imaging in assessing mucosal healing in patients with ulcerative colitis. Gastrointest Endosc. 2023 Apr;97(4):759-766.e1. doi: 10.1016/j.gie.2022.11.019. Epub 2022 Nov 30. PMID 36460084
- [Background] Neumann H, Vieth M, Gunther C, Neufert C, Kiesslich R, Grauer M, Atreya R, Neurath MF. Virtual chromoendoscopy for prediction of severity and disease extent in patients with inflammatory bowel disease: a randomized controlled study. Inflamm Bowel Dis. 2013 Aug;19(9):1935-42. doi: 10.1097/MIB.0b013e318290550e. PMID 23839228
- [Background] Pabla BS, Schwartz DA. Assessing Severity of Disease in Patients with Ulcerative Colitis. Gastroenterol Clin North Am. 2020 Dec;49(4):671-688. doi: 10.1016/j.gtc.2020.08.003. Epub 2020 Sep 23. PMID 33121688
- [Background] Katsanos KH, Papamichael K, Christodoulou DK, Cheifetz AS. Histological healing beyond endoscopic healing in ulcerative colitis: Shall we target the "ultra-deep" remission? Dig Liver Dis. 2017 Dec;49(12):1332-1333. doi: 10.1016/j.dld.2017.08.043. Epub 2017 Sep 18. No abstract available. PMID 28964677